CLINICAL TRIAL: NCT05931198
Title: Incorporation de prothèses Chez Les Patients amputés de Membre supérieur à l'IRMA
Brief Title: Several Studys Showed That Upper Limb Amputated Patients Are Able to Experience the Illusion of the Rubber Hand Whith Prosthesis: We Want to go Futher by Comparing the Strength of the Incorporation According to the Type of Prosthesis Using the Illusion of the Rubber Hand With Prothesis
Acronym: MYARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Robert Merle d'aubigné (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22.03801.000168
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Appropriate Affect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper limb amputee population (Experimental)
  Interventions: Other: Modified illusion of the rubber (syncrhone); Other: Modified illusion of the rubber (asynchrone)

INTERVENTIONS:
Other: Modified illusion of the rubber (syncrhone) — The residual limb of the patient will be hide for the patient. The prothesis and the other hand of the patient will be visible. The investigators are going to touch the residual limb and the prothesis at the same time (synchrone) during at least 2 min. The investigators will ask to the patient to point where they felt the touching spot on a tray with measurement grid and to asnwer to the pre-prepared questionnaire.
Other: Modified illusion of the rubber (asynchrone) — The residual limb of the patient will be hide for the patient. The prothesis and the other hand of the patient will be visible. The investigators are going to touch the residual limb and the prothesis not at the same time (asynchrone) during at least 2 min. The investigators will ask to the patient to point where they felt the touching spot on a tray with measurement grid and to asnwer to the pre-prepared questionnaire.

SUMMARY:
The goal of this observational study is to compare the strength of the incorporation according to the type of prosthesis (aesthetic, mechanical, myoelectric) with the experience the illusion of the rubber hand. The investigators will replace is the rubber by the patient's prothesis. The population will be people with upper arm amputation above the hand and they will be their own comparation.

Participants will do the the experience the illusion of the rubber hand in asynchronic and synchronic way and to answer questionnaries.

ELIGIBILITY:
Inclusion Criteria:

* At least one upper limb amputation
* Informed and consented to participate to the study

Exclusion Criteria:

* having a history of severe neurological, visual or musculoskeletal impairments (other than the loss of a limb)
* with severe serious psychiatric disorders (e.g. schizophrenia)
* having problems understanding French in order to guarantee a good understanding of the questionnaires
* under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Proprioceptive drift | Immediately after the intervention
  Before and after each intervention, we are going to ask to the patient to point where we touch the residual limb on a graduated board.

SECONDARY OUTCOMES:
Appropriate affect | Immediately after the intervention
  After each intervention, patient will answering to a questionnary about appropriation with their past as comparaison.
Influence of patient's characteristic | During the patient's inclusion / Baseline
  Compare patient's characteristic with other outome : amputation level, time since amputation, time using the prothestics

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Robert Merle d'Aubigné, Valenton, France

REFERENCES:
- [Background] Botvinick M, Cohen J. Rubber hands 'feel' touch that eyes see. Nature. 1998 Feb 19;391(6669):756. doi: 10.1038/35784. No abstract available. PMID 9486643
- [Background] Ehrsson HH, Rosen B, Stockselius A, Ragno C, Kohler P, Lundborg G. Upper limb amputees can be induced to experience a rubber hand as their own. Brain. 2008 Dec;131(Pt 12):3443-52. doi: 10.1093/brain/awn297. Epub 2008 Dec 11. PMID 19074189